CLINICAL TRIAL: NCT06664749
Title: Comparison of the Effects of Three Stair Positioning Pillows and Positioning Materials on the Sleep-Wakefulness Status of Preterm Infants
Brief Title: Sleep-wakefulness Status in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma BOZDAG, Associate Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HRU-BOZDAG-003
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sleep
Keywords: preterm; infants; neonatal intensive care unit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three stair position pillow group (Experimental): Three stair position pillows were used for preterm infants.
  Interventions: Other: Three stair position pillow group
- Positioning material group (Experimental): Positioning materials were used for preterm infants.
  Interventions: Other: Positioning material group

INTERVENTIONS:
Other: Three stair position pillow group — Preterm infants were monitored with three stair position pillows.
  Arms: Three stair position pillow group
Other: Positioning material group — Preterm infants were monitored with positioning material pillows.
  Arms: Positioning material group

SUMMARY:
This study was conducted to compare the effectiveness of three stair positioning pillows and positioning materials on the sleep-wakefulness status of preterm infants.

DETAILED DESCRIPTION:
It is known that newborns have similar brain activity in the intrauterine period and REM sleep activity, and they sleep more than adults and spend most of their sleep in the REM sleep period. Therefore, sleep quality in the newborn period is directly related to healthy development. Providing a developmentally supportive position in neonatal intensive care units (NICU) is necessary not only for neuromotor and musculoskeletal development, but also for physiological function and stability, thermal regulation, bone density, neurobehavioral organization, calmness and comfort, skin integrity, optimal musculoskeletal development, facilitation of sleep, growth and brain development. Excessive noise in the NICU, prolonged bright lights, separation from the mother, frequent invasive procedures and pain experience are among the factors that disrupt, shorten and create stress in the sleep duration of preterm babies. It is very important to support the sleep of preterm babies in the NICU in order to improve their growth and development, especially their brain development. It is known that therapeutic positions, which are one of the individualized developmental care practices, are effective on sleep.This study was conducted to compare the effectiveness of three stair positioning pillows and positioning materials on the sleep-wakefulness status of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants who were postmenstrual age ≥30 and ≤34,
* had an appropriate weight for gestational age (AGA),
* were spontaneously breathing (extubated and not receiving any oxygen support),
* had no history of previous intubation, routinely had caffeine in their diet, and
* whose parents volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Preterm infants who were <30 and >34 years postmenstrual,
* had bradycardia,
* received an analgesic 4 hours before that could affect sleep,
* had sepsis,
* congenital anomalies,
* intracranial hemorrhage,
* hyperbilirubinemia,
* hypoglycemia,
* underwent surgery,
* received any oxygen support, or were on mechanical ventilation were excluded from the study.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Sleep | 3 hours
  Measured with an actigraphy device. Unit is minutes.
wakefulness | 3 hours
  Measured with an actigraphy device. Unit is minutes.

CONTACTS AND LOCATIONS:
Overall Officials: fatma bozdağ, Principal Investigator — Harran University
Locations (1):
- Fatma Bozdağ, Sanliurfa, Turkey (Türkiye)